Evaluation of Lens Rotation in Habitual Wearers of Toric, Soft Contact Lenses

Protocol CR-6576

Version: 1.0

Date: 03 October 2024

#### Test Articles:

Marketed ACUVUE® OASYS 1-Day for Astigmatism contact lenses (Test Lens) from JJVCI and Dailies® Total1 for Astigmatism contact lenses (Control Lens) from Alcon Inc.

Commercially Available Product Lots: ACUVUE® OASYS 1-Day for Astigmatism contact lenses from JJVCI and Dailies® Total1 for Astigmatism contact lenses from Alcon Inc.

Keywords: Astigmatism, senofilcon A, ACUVUE® OASYS 1-Day for Astigmatism, Dailies® Total1 for Astigmatism contact lenses from Alcon, delefilcon A, daily wear, daily disposable, non-dispensing, Visual Analogue Scores, logMAR visual acuity, rotation performance.

### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This clinical trial will be conducted in compliance with ISO 14155:2020<sup>1</sup>, Declaration of Helsinki<sup>2</sup>, United States (US) Code of Federal Regulations (CFR)<sup>3</sup>, and International Council for Harmonization Good Clinical Practice E6(R2) (ICH GCP)<sup>4</sup>.

### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.









## PROTOCOL TITLE, NUMBER, VERSION AND DATE

Title: Evaluation of Lens Rotation in Habitual Wearers of Toric, Soft Contact Lenses

Protocol Number: CR-6576

Version: 1.0

Date: 03 October 2024

### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

### MEDICAL MONITOR



The Medical Monitor must be notified by the clinical institution/site by e-mail or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards the assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

### **AUTHORIZED SIGNATURES**

The signatures below constitute the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements, ISO 14155:2020, Declaration of Helsinki<sup>2</sup>, and the United States (US) Code of Federal Regulations (CFR)<sup>3</sup>, and International Council for Harmonization Good Clinical Practice E6(R2) (ICH GCP)<sup>4</sup>





# **SYNOPSIS**

| Protocol Title | Evaluation of Lens Rotation in Habitual Wearers of Toric, Soft Contact<br>Lenses |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Clinical trial phase: Feasibility |
| | Design control phase: Development phase, phase 0. |
| Trial Registration | This study will be registered on ClinicalTrials.gov by the sponsor. |
| Test Article(s) | Investigational Products: None |
| | Approved Products (locally sourced by research site): 1. ACUVUE® OASYS 1-Day for Astigmatism (AO1DfA) contact lenses for Johnson and Johnson Vision Inc. (Test Lens) 2. Dailies® Total1 for Astigmatism (DT1fA) contact lenses from Alcon Inc. (Control Lens) |
| Wear and Replacement | Wear Schedule: daily wear |
| Schedules | Replacement Schedule: daily disposable |
| Objectives | Primary Objective: |
| oojeenves | The primary objective of this study is to measure the monocular distance (6m) logMAR visual acuity with each study lens (Test lens and Control lens) after lens fitting. |
| | Other (Exploratory) Objectives: The exploratory objectives of this study include changes in lens orientation after settling and over time with an automated lens tracking system; VAS scores after lens fitting for vision, comfort and handling; and lens orientation at 1, 3, and 15-minutes following insertion. Adverse events and slit lamp findings will also be monitored and collected. |
| Study Endpoints | Primary Efficacy Endpoint: 1. Distance Visual Acuity |
| | <ol> <li>Other (Exploratory) Efficacy Endpoints: <ol> <li>Lens orientation measured over time with an automated lens tracking system following intentional misalignment</li> <li>Lens orientation recorded with an automated lens tracking system following eye movements</li> <li>Settling Time following intentional misalignment</li> <li>Toric Lens orientation at 1-, 3-, and 15-minutes following insertion</li> </ol> </li> <li>Subjective Vision, Comfort and Handling Scores approximately 15-minutes after lens insertion</li> </ol> |
| | Other Safety Endpoints: |
| | Adverse Events (AEs) |
| | 2. Slit Lamp Findings (SLFs) |

| | T=1 == 1 = 1 |
|---|---|
| Study Design | This will be a single site, 2-visit, randomized, controlled, single-masked, non-dispensing, bilateral wear, 2×2 cross-over study. Each subject will be randomly assigned to one of two wear sequences. There will be a washout period of 1-10 days in between the visits. There will be a total of 2 visits: |
| | Visit 1: Screening, baseline evaluation and lens fit #1 |
| | Visit 2: Continuance, lens fit #2, Exit evaluation |
| | See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (). |
| Sample Size | This study will have an enrollment target of approximately 7 subjects, with a target of at least 5 to complete. This is a crossover study, and all subjects will be randomized to one of 2 unique sequences of lens wear. |
| Study Duration | Total study duration including the enrollment period is anticipated to be approximately 6 weeks. The expected duration of participation of the subject will be approximately 1 week. |
| Anticipated Study Population | Subjects will be habitual toric, soft contact lens wearers with bilateral astigmatism who are between 18 and 39 years of age (inclusive). |
| Eligibility Criteria - Inclusion | Potential subjects must satisfy of all the following criteria to be enrolled in the study. |
| | Inclusion Criteria following Screening |
| | The subject must: |
| | <ol> <li>Read, understand, and sign the STATEMENT OF<br/>INFORMED CONSENT and receive a fully executed copy</li> </ol> |
| | of the form. 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol. |
| | <ol> <li>Be between 18 and 39 years of age (inclusive) at the time of</li> </ol> |
| | screening. 4. Habitually wear soft, toric contact lenses in both eyes in a |
| | daily or daily disposable wear modality (i.e. not extended |
| | wear modality). Habitual wearer is defined as a minimum of |
| | 6 hours per day, for a minimum of 2 days per week during |
| | the past 30 days. |
| | <ol> <li>Possess a wearable pair of spectacles that provide correction<br/>for distance vision (if applicable).</li> </ol> |
| | Inclusion Criteria at Baseline Evaluation |
| | The subject must: |
| | 6. Have the spherical component of their vertex-corrected distance refraction within the range +4.00 to -6.00 DS |
| | (inclusive) in both eyes. 7. Have the magnitude of the negative cylindrical component |
| | 7. Have the magnitude of the negative cylindrical component of their vertex-corrected distance refraction between 0.75 |
| | DC and 2.50 DC in both eyes. |
| | 8. Have best corrected monocular distance logMAR visual |
| | acuity of 0.2 or better in each eye. |

| BE THE CLU TO THE | In |
|---|---|
| Eligibility Criteria – Exclusion | Potential subjects who meet any of the following criteria will be excluded from participating in the study. |
| | Exclusion Criteria following Screening |
| | The subject must not: |
| | Be currently pregnant or lactating. |
| | 2. Be diabetic. |
| | 3. Be currently using any ocular medications or have any ocular |
| | infection of any type. |
| | <ol> <li>By self-report, have any ocular or systemic disease, allergies,</li> </ol> |
| | infection, or use of medication that might contraindicate or |
| | interfere with contact lens wear, or otherwise compromise study<br>endpoints, including infectious disease (e.g., hepatitis, |
| | tuberculosis), contagious immunosuppressive disease (e.g., |
| | Human Immunodeficiency Virus [HIV]), autoimmune disease |
| | (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of |
| | serious mental illness or seizures. See section 9.1 for additional |
| | details regarding excluded systemic medications. |
| | 5. Have habitually worn rigid gas permeable (RGP) lenses, |
| | orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, |
| | SoftPerm) within the past 6 months. 6. Be currently wearing monovision or multifocal contact lenses. |
| | 7. Be currently wearing lenses in an extended wear modality. |
| | 8. Be currently wearing or have had worn Acuvue® Oasys 1-Day for |
| | Astigmatism, or Dailies® Total1 for Astigmatism lenses during |
| | the last 3 months. |
| | 9. Have a history of strabismus or amblyopia. |
| | 10. Be an employee (e.g., Investigator, Coordinator, Technician) or |
| | immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee |
| | or their spouse) of the clinical site. |
| | 11. Have participated in a contact lens or lens care product clinical |
| | trial within 7 days prior to study enrollment. |
| | Exclusion Criteria at Baseline Evaluation |
| | The subject must not: 12. Have clinically significant (grade 3 or higher on the Efron |
| | grading scale) slit lamp findings (e.g., corneal edema, |
| | neovascularization or staining, tarsal abnormalities or bulbar |
| | injection) or other corneal or ocular disease or abnormalities that |
| | contraindicate contact lens wear or may otherwise compromise |
| | study endpoints (including entropion, ectropion, chalazia, |
| | recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis). |
| | 13. Have fluctuations in vision due to clinically significant dry eye or |
| | other ocular conditions. |
| | 14. Have had or have planned (within the study period) any ocular or |
| | intraocular surgery (e.g., radial keratotomy, PRK, LASIK, |
| D: 11 1 | iridotomy, retinal laser photocoagulation, etc.). |
| Disallowed Medications/Interventions | Subjects will not be eligible to enroll if they are taking any ocular |
| iviedications/interventions | medications, or any systemic medications that would normally contraindicate contact lens wear or may otherwise compromise study |
| | endpoints. See section 9.1 for details regarding disallowed systemic |
| | medications. |

| Measurements and Procedures Microbiology or Other | The key procedure associated with the primary endpoint for this study will be the evaluation of monocular logMAR visual acuity. Other measurements and procedures related to observational endpoints will include: - Lens orientation and stability in different time points following insertion - Lens rotation over time following intentional misalignment measured with an automated lens tracking instrument - Lens orientation following eye movements in 8 directions of gaze - Completion of the VAS questionnaires at fitting Not applicable for this study. |
|---|---|
| Laboratory Testing | |
| Study Termination | The occurrence of an Unanticipated Adverse Device Effect (UADE), Unanticipated Serious Adverse Device Effect (USADE), or Serious Adverse Event (SAE) for which a causal relationship to a test article cannot be ruled out, may result in stopping further dispensing of the test article. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | Non-preserved saline (locally sourced by research site) |
| Principal Investigator(s) and<br>Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept<br>separately from the Study Protocol and is included in the study Trial<br>Master File. |



### COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS

ADE Adverse Device Effect

ADHD Attention Deficit Hyperactivity Disorder
AE Adverse Event/Adverse Experience

AO1DfA ACUVUE OASYS® 1-DAY with HydraLuxe™ TECHNOLOGY for

ASTIGMATISM

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations

CI Confidence Interval

CLUE Contact Lens User Experience
COM Clinical Operations Manager
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

D Diopter

DMC Data Monitoring Committee
DT1fA Dailies® Total1 for Astigmatism
eCRF Electronic Case Report Form
EDC Electronic Data Capture
ESD Evelid Stabilized Design

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration GCP Good Clinical Practice HEV High Energy Visible

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus HLHC High-Luminance, High-Contrast

IB Investigator's Brochure

ICH The International Council for Harmonization

IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intention-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LASIK Laser-Assisted in Situ Keratomileusis

LogMAR Logarithm of Minimal Angle of Resolution

 OD
 Right Eye

 OS
 Left Eye

 OU
 Both Eyes

PIG Patient Instruction Guide
PQC Product Quality Complaint
PRK Photorefractive Keratectomy
PRO Patient Reported Outcome

QA Quality Assurance

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan
SAS Statistical Analysis System
SD Standard Deviation
SLF Slit Lamp Findings

UADE Unanticipated Adverse Device Effect
USADE Unanticipated Serious Adverse Device Effect

UV Ultraviolet
VA Visual Acuity
VAS Visual Analogue Scale

### 1. INTRODUCTION AND BACKGROUND

Johnson and Johnson Vision currently market ACUVUE® OASYS 1-Day for Astigmatism daily disposable contact lenses which uses Blink Stabilized Technology to achieve rotational stability, while other manufacturers use other prism or peri-ballast mechanisms for rotational stability.

This study is designed to assess monocular distance visual acuity with the two marketed study lenses. The study will also evaluate the rotational performance of the two marketed lenses using an automated lens tracking instrument and custom software developed by Eurolens Research, at the University of Manchester.



### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

### 2.1. Objectives

### **Primary Objective**

The primary objective of this study is to measure the monocular distance (6m) logMAR visual acuity with each study lens (Test lens and Control lens) after lens fitting.

### Other (Exploratory) Objectives

The exploratory objectives of this study include lens orientation and stability after settling, changes in lens orientation over time following intentional misalignment, changes in lens orientation following eye movements in 8 directions of gaze, VAS scores at fitting (comfort, vision, and handling), and lens orientation at 1- and 3-minutes following insertion. Adverse events will also be monitored and collected.

### 2.2. Endpoints

#### 2.2.1. Efficacy Endpoints

### **Primary Efficacy Endpoint**

1. Distance (6m) Visual Acuity

The primary endpoint for this study will be distance visual acuity measured monocularly at 6 meters after lens fitting under high-luminance high contrast (HLHC) lighting conditions using the Eurolens computerized logMAR VA chart. The logMAR VA score is a continuous endpoint.

#### Other (Exploratory) Efficacy Endpoints

### Lens orientation measured over time with an automated lens tracking system following intentional misalignment

Each study lens will be rotated in the temporal direction from its original position to its worst case orientation (90° from its settled position for the AO1DfA lens which has a bidirectional stabilization design, and 180° from its settled position for the DT1fA lens which has a unidirectional stabilization design), followed by video capture of the lens orientation over a 5-minute period. Lens orientation data (rotation error magnitude and direction relative to the 6 o'clock position, and rotation error magnitude and direction relative to original settled position) will be calculated at 5-second increments through the measurement period. Rotation error magnitude will be recorded in degrees (0 to 180), and rotation error direction will be recorded as base temporal or nasal. For the DT1fA lens type, recovery from 90° misalignment will also be determined from the timepoint that it reaches this position during the recovery from 180° of misalignment.

### 2. Lens orientation recorded with an automated lens tracking system following eye movements

Lens settled orientation (rotation error magnitude and direction relative to the 6 o'clock position) in primary gaze will be measured. Lens orientation will then be measured again after the subject has been asked to perform an eye movement in each of the eight cardinal directions of gaze. The difference in orientation (magnitude and direction) from before eye movement to after eye movement will be determined.

### 3. Settling Time following intentional misalignment

The time (in seconds) required for the study lenses to settle (defined as returning to within 5 degrees of initial settled position) after intentional misalignment will be recorded for each eye and lens during the assessment of the lens orientation recorded with an automated lens tracking system (Other efficacy endpoint 1). Settling time is a continuous endpoint.

### 4. Toric lens orientation

Toric lens orientation (scribe mark position relative to 6 o'clock) will be assessed for each eye at 1, 3 and at least 15 minutes after lens insertion at the fitting visit. The endpoint is the distribution (counts, percentages) of eyes for the toric orientation (in degrees). Toric lens stability with blink at least 15 minutes after lens insertion will also be recorded. See in Appendix D for details regarding the collection of lens orientation.

### 5. Subjective Vision, Comfort and Handling Scores

Vision, comfort and handling will be assessed monocularly approximately 15-minutes after lens insertion using individual questionnaire items with a Visual Analogue Scale (VAS). The VAS scale for each item is continuous set where scores range from 0 (represent worst imaginable vision, comfort, or extreme difficulty in lens handling) to 100 (represent best imaginable vision, comfort, or easiest to handle). Vision, comfort, and handling scores are continuous endpoints. See appendix A for the details of the study questionnaire.

### 2.2.2. Safety Endpoints

Primary Safety Endpoint Not applicable

Secondary Safety Endpoint Not applicable

### Other Safety Endpoint

- Adverse events (AEs) including ocular and non-ocular. Details for AEs will be provided through listings.
- Slit lamp findings (SLFs) the SLF grades determined using the Efron Grading Scale will be summarized descriptively.

#### 2.3. Hypotheses

Not applicable, no statistical hypothesis testing will be performed for any endpoints in this study.

### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

The target population for this study will be healthy adult soft, toric contact lens wearers between 18 and 39 years of age with binocular astigmatism.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

Inclusion Criteria following Screening

The subject must:

- Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- Be between 18 and 39 years of age (inclusive) at the time of screening.
- 4. Habitually wear soft, toric contact lenses in both eyes in a daily or daily disposable wear modality (i.e. not extended wear modality). Habitual wearer is defined as a minimum of 6 hours per day, for a minimum of 2 days per week during the past 30 days.
- Possess a wearable pair of spectacles that provide correction for distance vision (if applicable).

### Inclusion Criteria at Baseline Evaluation

The subject must:

- Have the spherical component of their vertex-corrected distance refraction within the range +4.00 to -6.00 DS (inclusive) in both eyes.
- Have the magnitude of the cylindrical component of their vertex-corrected distance refraction between 0.75 DC and 2.50 DC in both eyes.
- Have best corrected monocular distance visual acuity of 0.2 or better in each eye.

### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria following Screening

The subject must not:

- Be currently pregnant or lactating.
- Be diabetic.
- Be currently using any ocular medications or have any ocular infection of any type.
- By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that
  might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints,
  including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease

- (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
- Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
- Be currently wearing monovision or multifocal contact lenses.
- Be currently wearing lenses in an extended wear modality.
- Be currently wearing or have had worn Acuvue<sup>®</sup> Oasys 1-Day for Astigmatism, or Dailies<sup>®</sup> Total1 for Astigmatism lenses during the last 3 months.
- Have a history of strabismus or amblyopia.
- Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
- Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.

## Exclusion Criteria at Baseline Evaluation

The subject must not:

- 12. Have clinically significant (grade 3 or higher on the Efron grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
- Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
- Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

### 4. STUDY DESIGN AND RATIONALE

## 4.1. Description of Study Design

This will be a single site, 2-visit, randomized, controlled, single-masked, non-dispensing, bilateral wear, 2×2 cross-over study. Each subject will be randomly assigned to one of two wear sequences (AO1DfA followed by DT1fA or DT1fA followed by AO1DfA), with a 1-to-10 day(s) washout period between wear periods. Lens rotation will be assessed over time with a slit lamp as well as with an automated lens tracking software. Subjective comfort, vision and handling will be assessed using the VAS questionnaire at fitting for each wear period. High Luminance High Contrast LogMAR VA will be assessed. Subjects will not have access to the study lenses following completion of the protocol.

### 4.3. Enrollment Target and Study Duration

This study will have an enrollment target of approximately 7 subjects, with a target of at least 5 to complete. The study will be conducted at 1 clinical site. A subject will be considered enrolled upon signing of the informed consent form.

There will be 2 visits in total per subject; total study duration including the enrollment period is expected to be approximately 6 weeks. Subjects who are discontinued prior to the final evaluation may be replaced at the discretion of the study sponsor. The investigation will end at the time when all visits have been completed for all enrolled subjects and the study data is locked.

### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn bilaterally in a randomized fashion using a  $2\times2$  crossover design.

A computer-generated randomization scheme will be used to randomly assign subjects to one of two unique sequences of lens wear (AO1DfA/DT1fA or DT1fA/AO1DfA) using an allocation ratio of 1:1 between lens sequences.

The randomized assignment of subjects will be performed at the first visit prior to the first fitting. The Clinical site will follow the randomization scheme provided and will not pre-select or assign subjects. The following must have occurred prior to randomization:

- Informed consent must have been obtained
- The subject must have met all inclusion and exclusion criteria
- The subject history and baseline information must have been collected



### 5.2. Masking

This is a single-masked trial. Subjects will be masked to both study lenses. The study staff responsible for choosing the appropriate lens (site investigators or other site personnel) as per the randomization scheme will remove the foil from the packaging prior to providing lenses to subjects for lens insertion, so that the subjects may remain masked throughout the study.

Investigators and site personnel will not be masked to the study lenses due to the difference in packaging and lens markings.

#### 5.3. Procedures for Maintaining and Breaking the Masking

Not applicable. As this is a non-dispensing trial, there is no foreseen situation in which the site would need to inform the subject of what contact lens they are wearing.

### 6. STUDY INTERVENTION

### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Acuvue <sup>®</sup> Oasys 1-Day for<br>Astigmatism (Test) | Dailies® Total 1 for Astigmatism<br>(Control) |
|---|---|---|
| Test Article Form | Soft toric contact lenses | |
| Description | Standard marketed lenses | |
| Manufacturer | Johnson & Johnson Vision Care,<br>Inc. | Alcon Inc. |
| Packaging Form | Blister packaging with sterile packing solution | Blister packaging with sterile<br>packing solution |
| Packaging Solution | Optimized Borate Buffer (OBB)<br>solution | Packaged in solution containing wetting agents |
| Lens Material | senofilcon A | delefilcon A |
| Sphere Powers (DS) | Marketed SKUs (+4.00 to -6.00) | |
| Cylinder Powers (DC) | Marketed SKUs (0.75 to 2.50) | |
| Cylinder Axes (°) | Marketed SKUs | |
| Nominal Water Content (%) | 41 | Variable |
| Nominal Base Curve (mm) | 8.5 | 8.6 |
| Lens Diameter (mm) | 14.3 | 14.5 |
| Fiducial marks | 6 and 12 o'clock fiducial lines | 6 o'clock fiducial line |
| Dk | 103 | 140 |
| Wear Modality in Current<br>Study | Daily wear | |
| Replacement Frequency in<br>Current Study | Daily disposable | |
| Commercially available | Yes | Yes |

The site will be acquiring and using the commercially available lots to match the prescription per subject.

### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Non-Preserved Saline |
|------------------|-----------------------------------|
| Solution | Astroplast Ultra Saline 20ml Pods |
| Name/Description | or similar |
| Manufacturer | Wallace Cameron International Ltd |
| Preservative | None |

The sites will be acquiring the ancillary supplies as needed for the study including lens cases or fluorescein strips.

### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, for in-office wear only as part of the requirements set forth in this clinical protocol.























### 8. SUBJECTS COMPLETION/WITHDRAWAL

### 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent.
- they are eligible.
- have not withdrawn/discontinued from the study for any reason described in section.
- completed all visits through the final visit (Visit 2).
- If all visits were completed but an additional visit is considered necessary for subject care, follow the requirements for unscheduled visits in section.

### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject withdrawal of consent.
- · Subject not compliant to protocol
- Subject lost to follow-up.
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant).
- Subject develops significant or serious adverse events necessitating discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE).
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment).
- Subject missed any study visits
- · Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort
  or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled).
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- · Record the spherocylindrical refraction with best corrected distance visual acuity.
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless
  otherwise stated in section 7.2.
- Collect all unused test article(s) from the subject.
- Make arrangements for subject care, if needed, due to their study participation

Additional subjects may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed concomitant interventions for this study include ocular medications of any kind, or any systemic medications that would normally contraindicate contact lens wear or may otherwise compromise study endpoints.

#### 9.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film.

A summary of disallowed systemic medications is shown in . Subjects with a history of taking these medications will be allowed to enroll only if:

- The medications have been taken on a continual, routine basis for at least 6 months, and
- The subject has demonstrated successful contact lens wear during this time.

Or:

The subject was taking the medication on a temporary basis and ceased taking that medication at least 2
weeks prior to signing the informed consent (this is considered sufficient time for the medication to have
left the body prior to enrollment).

Subjects with a history of taking medications listed in on a long-term, routine basis for less than 6 months will not be allowed to participate in the study.

Table 4: Disallowed systemic medications

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Estrogens (not including contraceptive medication) | Menopause, osteoporosis, vaginitis | Vagifem, Estrace, Climara, Vivelle-Dot, Premarin, Minivelle, etc. |
| Anticholinergics | Irritable bowel syndrome, Parkinson's disease, peptic ulcer, cystitis, nasal congestion, cold symptoms, overactive bladder, COPD | Bentyl, Spiriva, Atrovent, Hyosyne,<br>Levsin, Symax Fastab, Symax SL,<br>Homax SL, Cogentin, Transderm Scop,<br>etc. |
| Beta-blockers | Hypertension, angina, heart attack,<br>migraine, atrial fibrillation, adrenal<br>cancer, essential tumor, glaucoma | Toprol XL, Lopressor, Tenormin,<br>Propranolol, Timoptic, Trandate, Inderal<br>LA, etc. |
| Psychotropics | Antipsychotic (schizophrenia, mania),<br>antidepression, antiobsessive, antianxiety,<br>mood stabilizer, stimulants (ADHD) | Zoloft, Celexa, Prozac, Lexapro,<br>Effexor, Cymbalta, Ativan, Xanax,<br>Desyrel, Wellbutrin, etc. |
| Vitamin A analogs | Cystic acne | Isotretinoin |

Examples of disallowed systemic antihistamines are given in . Subjects with a history of taking systemic antihistamines will be allowed to enroll only if:

- They have taken antihistamines continuously for at least 2 weeks, and
- · They have demonstrated successful wear while taking the medication

Or:

• They stopped taking the medication for at least 2 weeks prior to enrollment.

Table 5: Disallowed systemic antihistamines

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Antihistamines | Allergic rhinitis, sedation, hives, allergic conjunctivitis, skin allergy, itching, motion sickness | |

### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, to the IEC/IRB.

If the deviation potentially impacts the safety of subject or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation". Deviations that contradict the information contained in the Informed Consent/Assent forms will be considered Major Deviations.

Minor deviations have no substantive effect on subject safety or technical integrity of the study. They are often logistical in nature.

Protocol waivers are prohibited.

lists examples of deviations that will constitute major and minor protocol deviations for this study.

Table 6: Examples of major and minor protocol deviations

| Deviation category | Major deviation | Minor deviation |
|---|---|---|
| Out-of-window visit (applies to<br>wear periods only, i.e. not washout<br>period) | Visit attended > 2 days out of visit<br>window defined in study<br>procedures | Visit attended ≤ 2 days out of visit window defined in study procedures |

In the case of a major protocol deviation, the decision of whether or not the subject will be excluded from the Per-Protocol analysis population will be made at the time of cohort review. The list of major deviations with potential impact on the primary endpoint will be flagged separately and used to define the per protocol population.

#### 11. STUDY TERMINATION

If more than 2 subjects in the investigational soft contact lens group develop serious expected (e.g., definite or probable MK) or unexpected device related adverse events, the study will be suspended. Upon review and consultation with IRB, DMC, and JJVC Safety Management Team, the study may be terminated. This potential stopping rule is established based on our trial involving approximately 200 subjects wearing the investigational soft contact lens for up to 3 years with an assumed MK rate that is below 0.2% per subject-year. The rate of 0.2% per subject-year is the established rate for extended wear lenses in adults, which was requested by the FDA as a criterion for evaluating a contact lens for pediatric use in an FDA response to a pre-IDE submission. To be conservative, 200 independent subject years were used in the calculation. The probability of observing 2 cases or

more incidents of MK is 0.061, and 3 cases or more incidents of MK is 0.007 (given an MK rate of 0.2% per subject year).

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on subject safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason and will follow the internal applicable quality review process and will notify the IEC/IRB. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness, or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff caused by handling by the user, and not indicative of a
  quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the
  subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).

- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.
- Confirmation of product availability for return (and tracking information, if available), or rationale if
  product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also apply and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

Adverse Event (AE) – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated."

NOTE: This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- Was not present prior to the study, but appeared or reappeared following initiation of the study.
- Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.

NOTE: Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) - An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
  - Life-threatening illness or injury
  - Permanent or persistent impairment of a body structure or a body function
  - Hospitalization or prolongation of patient hospitalization
  - Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
  - Chronic disease
- Foetal distress, foetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization

- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

Significant Adverse Events – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related comeal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Hordeolum
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks</li>

Adverse Device Effect (ADE) – An ADE is an "adverse event related to the use of an investigational medical device."

NOTE 1: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

NOTE 2: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.

NOTE 3: This includes 'comparator' if the comparator is a medical device.

Serious Adverse Device Effect (SADE) - Any adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.

**Unanticipated Serious Adverse Device Effect (USADE):** serious adverse device effect (SADE) which by its nature, incidence, severity or outcome has not been identified in the current risk assessment. [USADE is synonymous with UADE below from the United States (US) Code of Federal Regulations (CFR)<sup>3</sup>.]

NOTE 1: Anticipated serious adverse device effect (ASADE) is an effect which by its nature, incidence, severity or outcome has been identified in the risk assessment.
Unanticipated Adverse Device Effect (UADE) – A UADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects. [UADE is synonymous with USADE above from ISO 14155<sup>1</sup>.]

### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study
  procedures and the adverse event (not related, unlikely related, possibly related, or related)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse
  event (mild, moderate, or severe)
- Outcome not recovered or not resolved, recovering or resolving, recovered or resolved with sequelae, recovered or resolved, death related to adverse event, or unknown.
- Actions Taken none, temporarily discontinued, permanently discontinued, or other.

### Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article, study treatment, or the study procedures. The test article, study treatment, or study procedures relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment, or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug)
  and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of
  concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge
  and re-challenge.

### Severity Assessment

Severity Assessment – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's
  daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs and complete the Adverse Event eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted (where appropriate), including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if the AE is related to the visual system.

Upon discovery of an AE that is deemed 'possibly related' or 'related' to the test article or study procedures (whether related to the visual system or not), an AE review form must be completed. Additional dated and initialed entries should be made at follow-up evaluations. Separate forms must be completed for each eye if the AE is bilateral.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the subject will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events

that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by EDC System, e-mail, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements. The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

### Reporting Adverse Events to Sponsor

### Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by EDC System, e-mail or, telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event
  was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

### Unanticipated (Serious) Adverse Device Effect (UADE)

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

### Non-Serious Adverse Events

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

### Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according to the written guidelines, including reporting timelines.

### 13.5. Event of Special Interest

None

### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant subject and their fetuses will not be monitored for study related purposes. Pregnant subjects are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

### 14. STATISTICAL METHODS

### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

Descriptive summary tables (descriptive statistics and/or frequency tables) will be provided for all demographic and baseline characteristics, efficacy variables and safety variables. For continuous endpoints, the descriptive statistics will include the number of subjects and/or eyes (as appropriate), mean, standard deviation (SD), median, and minimum and maximum. For binary or categorical endpoints, the frequency distribution with the number and percentage of subjects and/or eyes (as appropriate) in each category will be calculated. Graphic displays may also be used to summarize the data. Unscheduled visits will be summarized separately.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC)<sup>5</sup>.

### 14.2. Sample Size Justification

This study was not designed or powered to test any statistical hypotheses with respect to distance (4m) visual acuity. As this will be the first study that will utilize the tracking software (Open Source Physics – OSP) a total of 5 subjects (10 eyes) to complete the study was based on clinical considerations and operational feasibility. A total of 5 subjects under a 2×2 crossover design provides sufficient data to evaluate the efficiency of this new software.

### 14.3. Analysis Populations

### Intention-to-Treat (ITT) Population:

Intention-to-treat population will include all randomized subjects. Subjects will be analyzed as per planned randomized treatment.

### Safety Population:

All subjects who are administered any study intervention. Subjects will be analyzed as per actual treatment received.

### Per-Protocol Population:

All subjects who successfully complete all visits and do not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock. Justification for the exclusion of subjects with protocol deviations from the per-protocol population set will be documented in a memo to file.

### 14.4. Level of Statistical Significance

Not applicable. No hypothesis testing will be performed for any endpoints in this study.

### 14.5. Statistical Analyses

### Handling of Missing Data

All data summaries and statistical analysis will be conducted using the observed case data without multiple imputation. The count of missing data will be provided in each listing and table provided.

### 14.6. Efficacy Analyses

All efficacy endpoints will be summarized for both the ITT and per-protocol population using observed case data without multiple imputation.

### **Primary Efficacy Endpoint**

### Distance Visual Acuity

Distance (6m) monocular HLHC logMAR visual acuity at fitting will be summarized and presented only descriptively by lens type and timepoint (if applicable). Summary statistics are described in section 14.1

### Secondary Efficacy Endpoint

Not applicable.

### Other Efficacy Endpoints

- 1. Lens orientation measured over time with an automated lens tracking system following intentional misalignment Data resulting from the processing of the videos of each subject eye (for each lens), will be summarized by parameter (rotation error magnitude [range: 0 to 180] and rotation error direction [base temporal or nasal]). The video processed will be approximately 5 minutes per eye per lens. The tracking software will measure the parameters at 5-second intervals, totaling for a plan of 60 observations per eye per lens. Rotation error magnitude is a continuous data point while the rotation error direction is nominal categorical data. Signed rotation will be derived based on rotation error magnitude and direction and will be included as part of the external data file detailed in section 15. Parameter data (rotation error magnitude, signed rotation, and rotation direction) reported (or derived) from the automated tracking system will be summarized as per section 14.1.
- 2. Lens orientation recorded with an automated lens tracking system following eye movements
  In addition to collecting rotation error magnitude and direction following intentional misalignment,
  rotation error magnitude and direction will be recorded in each of the 8 cardinal gaze directions before
  and after eye movement. The singed rotation will be derived in the same manner as described above.
  Summaries will be provided for each parameter (rotation error magnitude, singed rotation, and rotation
  direction), timepoint (before and after eye movement) and gaze separately. Additional summaries will
  be provided for the 8 gazes combined.

The 8 cardinal gazes are:

- Up and to the right
- Upward
- Up and to the left
- Right
- Left
- Down and to the right
- Downward
- Down and to the left

### 3. Settling Time following intentional misalignment

The time (in seconds) required for the lens to settle (defined as returning to within 5 degrees of initial settled position) after intentional misalignment will be presented descriptively and summarized separately for each study lens. Summary statistics are described in section 14.1.

### 4. Toric Lens Orientation

The distribution (counts, percentages) of eyes for the toric Orientation (in degrees) at 1- and 3-minutes after lens insertion will be summarized at fitting and by lens type. Summary statistics are described in section 14.1.

### 5. Subjective Vision, Comfort and Handling Scores

Vision, comfort, and handling items will be summarized separately and presented only descriptively by lens type and timepoint (if applicable). Summary statistics are described in section 14.1.

### 14.7. Safety Analyses

All safety endpoints will be summarized for the safety population using observed case data.

### **Primary Safety Endpoint**

Not applicable.

### Secondary Safety Endpoint

Not applicable.

### Other Safety Endpoints

### 1. Slit Lamp Findings

Slit Lamp Findings (SLF) related to study lens wear will be assessed for each eye at all study visits (scheduled and unscheduled). SLFs will be evaluated and graded using the Efron Grading scale. The Efron grading scale is interval continuous from 0 to 4, where 0 represents the absence of findings and findings > 0 representing successively worse findings. Slit lamp will be used to assess the following:

- Corneal infiltrates
- Conjunctival redness
- Limbal redness
- Corneal neovascularization
- Epithelial microcysts
- Corneal oedema
- Corneal staining
- Location of staining
- Conjunctival staining
- Blepharitis
- Meibomian Gland dysfunction
- Mucin ball

Each study lens and parameter will be summarized separately and presented descriptively.

### Adverse events (AEs)

Details for AEs will be provided through listings. This listing will include both ocular and non-ocular.

### 14.8. Interim Analyses

Not applicable.

### 14.9. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using a Sitero EDC system. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External data sources for this study include: Video files and Excel data files for lens orientation analysis per subject. Each video recording will show a single eye and its surrounding eyelid area (see Appendix G for example) without having personally identifiable information in the image or the filename. The video files will be provided in a standard video format (eg. mpeg). Video files are processed using tracking software (Open Source Physics – OSP) to estimate the lens orientation over a 5-minute period of recovery from intentional misalignment from the settled position. The rotation error direction and magnitude relative to two reference positions (relative to 6 o'clock position, and relative to initial settled position) will be provided. The signed rotation will be derived using rotation error magnitude and direction. Data is planned to be provided at 5 second increments, but alternative increments may be found to be necessary once data collection commences.

Additionally, lens orientation (direction and magnitude of rotation error relative to 6 o'clock position, and relative to initial settled position) following eye movements in 8 directions of gaze will be provided in a separate Excel spreadsheet.



authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2020.1

### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- · test article receipt/dispensing/return records
- date of study completion

reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

### 15.3. Trial Registration on ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov by the sponsor.

### 16. DATA MANAGEMENT

### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, including the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

### 16.4. Data Monitoring Committee (DMC)

Not applicable

### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

### 18. ETHICAL AND REGULATORY ASPECTS

### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study, and during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Subjects will only be enrolled if the subject is fully able to understand the risks, benefits, and potential adverse events of the study and provide their consent voluntarily.

### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, according to ISO 14155:2020, and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64th WMA General Assembly 2013<sup>2</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with applicable regulatory requirements.

### 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts
  of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- · If applicable, new or revised subject recruitment materials approved by the Sponsor
- · Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according
  to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- · Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

### 18.4. Informed Consent

Each subject, or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki, <sup>2</sup> and ISO 14155:2020<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subjects the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw their consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible
  with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- · accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

### 19. STUDY RECORD RETENTION

In compliance with the ISO 14155:2020, <sup>1</sup> guidelines, the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ISO 14155:2020, <sup>1</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports.

If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- · Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

### 21. PUBLICATION

The study will be listed on clinicaltrials.gov.











# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

- ACUVUE® OASYS 1-Day for Astigmatism contact lenses from JJVCI
   Dailies® Total1 for Astigmatism contact lenses from Alcon Inc.

measure destination for all supervised in a specificial trial frame to measure or estimate the "deft angle" of the options are in the supervised to the options are in comparate for the "deft" measure or estimate the "deft", then add or authoral it is comparate for the "deft", measure or estimate the "deft", then add or authoral it is no comparate for the "deft", the "deft is obtained to determine which deviction to compensate.

3. Trial Lens Fitting

The latter First per controlled by the wide of the first period or controlled by the

We must alway complete that maniporal results are studied in the mediate and individual and an advanced and a studied in the mediate and a spheropolated one reduction with a proposal series and a spheropolated convention from a correct series and the mediate former and the contract series and the media temporal learned formers are the correct series and the mediate former and a contract series and the mediate formers and the contract series and the contract series and the contract series are series and the contract series are series and the contract series are series and the contract and the contract series are series and an advanced as the contract series are the series and an advanced and as a series are series and an advanced and as a series are series and as a series and an advanced and a series are series and an advanced and a series are series and a series and an advanced and a series are series and an advanced and an advanced and an advanced and as a series are series and an advanced and an advanced and as a series are series and an advanced an advanced and an advanced and as a series and a series and an advanced and an advanced and an advanced and as a series and an advanced and an advanced and an advanced and as a series and an advanced an advanced and advanced an advanced and advanced and advanced and advanced and advanced and advanced

Compared and the compared and the compar

6. Other Supportions

5. Other Supportions

1. Other Supportions

PATIENT MANAGEMENT

The first is the restriction of the construction of the construction of the first is the construction of t

Nat (950) make the park in orders right from the 6 citical position by (7) and remosa stakes in the policy and content stakes in the policy of Corporate from the Corporation of Corporate from the Corporation of Section 1500 (200) and the

MULTIFOCAL FITTING GUIDELINES

2. Different particulars, and with the different particular of the work of the particular of the parti and and of and the man depth of any present service fresh contractions and for point rubes conquented to the point rubes construction and for point rubes construction to the point rube of any service in the point rubes contraction to the point rube

The first plane.

The first plane of the first plan WEARING SCHEDULE
he wanting achouse should be determined by the Eye Care Protessional Regular
hockupe, as determined by the Eye Care Protessional, are also orderenely important.

However, the parameters of the

asse Prescribed for they represent Replacement: energized for daily wear (frequent replacement), it is recommended that the be discorated and replaced with a new less early? Sweetic However, the Eye before and they determine an appropriate replacement achievable businesses responses of the palent.

4. Allow the larines to sotile for a minimum 10 minutes.
5. Assess places and then visitorizely and minutesculps.
6. Assess places are all we will conclude year throughout the second places and the places. All the source and an extra conclude and the second and

The characters was were stated delicated place, to then strike count on a considerable charge the construction of the charge of

Vasually demonstrate absolute to accord to a revoked during the initial resorting period. A profer may all first represence areas of branch size of Consects in Mandachies, and profer all personal represence and professional agreement in a sixeling of a sight inhaltoners for first all explaint his additional agreement between professional agreement in the programment of the cold in these or several independence. The largest these agreement is programed for according disagration.

When between an disposalte to the Contribution of the Contribution

is recommended that the contact liers wearer first be evaluated on a daily wear chockle. If successful, then a gradual introduction of entended wear can be followed a elemined by the prescribing Eye Care Professional. milmed by the prescritoring by the remreasors.

We display the prescritoring by the remreasors.

We display diseise can achieve the maximum west time.

Therspectic less west, does supervision by the fig. Che Protessional is noon

the more can be worn if received west for up to 6 ingitals of supervisional in the common for the common f

In this life is magniturious our selector that are since the face are be known in a contribulate lumine reservent card as in the horns.

Son patients that account card as in the horns.

For adjustment that account of the patient of the operation of the adjustment of the objection of the patients of most of the patients of most of the patients of th

A Patent Selection
Monosities deseale Assessment
A group programie, the patent should be selected distance and near
visual such in each pasent should have adequately corrected distance and near
visual such in each see, the armbyogic patent with significant amounts of incrommodal
adegrateful greater than 1,000 in one spe may not be a good candidate for moronicis
control and these times.

conservance unrest unest and security and a plant in considered, If the patient Occapions and experimental and demonsh should be considered. If the patient where the patient on include and patients are considered to the construction of the construction of the security of the construction and the experimental designment and the experimental design and the construction and the construction of the construction of the patients of the construction of the constructi

All plants in our floatest appeal and instructions to plant may not be present as an effect occurred to the control of the plants and the control of the plants and the control of the plants and the control of the plants and the plants and the plants and the plants and the plants are all the plants and the plants and the plants are all the plants are all the under a plant are all the plants are all the under a plant are all the may also the the control of the trans view. The blants are all the plants are all the under a plant are all

Con starth term it applicat in a life assist plants; package containing buffered staff

\* ADMIC BUSINES has core, power, downwise it marries, and expense of

\* ADMIC BUSINES has core, power, downwise it marries, and expense of

\* ADMIC BUSINES has core, power, downwise it marries, and expense of

\* ADMIC BUSINES has core, power, downwise, opficier,

\* ADMIC BUSINES AND THE PRESS PURPLE, base core, power, damenter, opficier,

and septimized feet.



Outbroom & Johnson Case, Inc. 2023

Read Advisors (Johnson & Johnson (Jonala) Inc.
In LSA, Johnson & Johnson Visin Case Inc.
Printed in USA
SAP Part Natures 2002/135
Revision Date (2020/235
Revision Naturber: A04.02.23-05

In 1 God of Portions Designation Methods the hope of t

Country probablish to be left also of the doke will burstler best with the A neutral probablish country to be left also of the doke will burstler best with the Country for the country of the country of the country of the country of the Library Country of the country of the

PACKAGE INSERT & FITTING INSTRUCTION GUIDE

ACUVUE QASYS

ACUVUE OASYS® Brand Contact Lenses ACUVUE OASYS® Brand Contact Lenses for PRESBYOP/ ACUVUE OASYS® Brand Contact Lenses for PRESBYOP/U WITH HYDRACLEAR® PLUS

senofilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily and Extended Wear

IMPORTANT: Please read carefully and keep this information for future use.

This Poskago Insett and Efficia Guide is infended for the Eye Care Protessional, ast advant in sense available to publish to proportion.

The Eye Care Protessional should proport in The Eye Care Protessional should provide the patient with the appropriate instructions that persists to the publish or pracected intenset. Copies are available for developed at seven-screen con-

RONN CAUTON U.S. Federal law restricts this device to on the order of a licensed practitioner. JJVC CONFIDENTIAL



| And a second that contact from waters who are amoleus have a highor ocidence of adverse resistors than recentions. We will not a second the contact from the control of the contact from the contact from the control of the control o |
|---|
|---|

# we are pleased independent of the control of the process on and care of control times in composition to control on the control of the control

when the throughous that has the series which wish one or or listenes liven in how me more and me was referred in our system. It was so that the best of the control of the control of the control of the desirable for and then not epicies have made as so part like for the helicensed should be control to the recommendation regardly swaring listenes charge any activity inches water. It is commendation regardly swaring listenes charge any activity inches water. As so they are Showing by the Lineae

Use of the must jurpose (cortact lene desidecting solution such time the lene seroakel (secret).

Water sould present,

Water sould present,

Do instructor or good for desident bit the lene cause since solution reuse evolution.

Do instructor or good for desident in the lene cause and control or

Discount that an Marki-Paper Schielen Bettle
Discount that an Marki-Paper Schielen Bettle
Discount to you making to show the the recommonds law prior included
Distort to you making to show on the to recommission to the bettle former on the to districtly and resident to the bettle make and by appear end to count to districtly and resident the
Contact bettle and the paper on the to the tent of countries and the country
are not provided the bettle bettle bettle bettle product to an elde use for any any experience of the countries of the paper of th

WARNING: Using multi-purpose solution beyond the discard date could result in c the solution and can lead to sewire infection, vision loss, or blindness,

CR-6576, v 1.0 20602135\_ACUVUE\_Oasys\_Hydrack

| )> | Lens Orientation Correct |
|---|---|
| have shown that contact lens wearers w<br>e of adverse reactions than nonsmokers | are shown that contact lons wearers who are smokers have a higher of arberese reactions than nonsmokers. |
| ith contact lenses ( | with contact lenses or lens care products could result in serious injury to<br>Patients should be curtificined that proceer use and care of contact lenses and |

Land continuidos, (20 NOT text) the of centaries in any softwar. Applica capital and the continues.

• the hast afficient times the centaries, (20 NOT text) to other bettless or centaries.

• the hast afficient times
in consistent the centaries the point design on any leaves to be subject to the centaries of the centering of the centaries of the centering of th

Circy and descount are come with described point with which deficiently of address country and control and a contr

Contract DAY

C 

Package Opening Icon (Blister)

图,智

MD

EC REP

14.0 mm Minus Lens - varies with power (e.g. -4.000: 0.070 mm) Plus Lens - varies with power (e.g. +4.000: 0.168 mm)

The procession of the processi In page design that of the other can be paged to consider the other can be a second or consider that the can be a second or can

TRANSMITTANCE CURVE 8.4 mm, 8.8 mm – 100 to e. 600 (e. 1020 interements) 4.5 00 to -12.000 (ei 0.200 interements) 4.5 00 to -12.000 (ei 0.200 interements) 4.5 00 to -8.000 (ei 0.500 interements) – 4.5 00 to -8.000 (ei 0.500 interements) – 20 mm to v. 87/104/1018 as to immigratical shelle of

ACUVIC OASYS

(seedfoord A)

(seedfoord A)

(seed Contact Lens

For Myopia'

24 YR, CUD

HUMAN CORNEAN

---- 25 YR, CUD HUMAN

CRYSTALLINE LENS? 8.6 mm plans 6.000 (a.020) incremental 4.020 to 4.000 (a.020) incremental 4.020 to 4.000 (a.020) incremental (plane, 1.020, 1.020, 1.250, 2.730 beau (\*\* 1.020) in (\*\* 2.730, 2.730 hear (\*\* 1.020) in (\*\* 2.730, 2.730 2.7401, Leone for \*\* 1.020) in (\*\* 2.730) in (\*\* 2.730)

Minus Lens - varies with power (e.g. -4.000: 0.080 mm) Plus Lens - varies with power (e.g. +4.000: 0.172 mm)

Base Curve (BC): Powers (D):

The ACUNUE DASYS® Brand Con the following dimensions: Diameter (DIA): Center Thickness: The data was debated two measurements below forced the coreal's 5 mm porters for the beneat morehold best 1,5 mm porters for the beneath terror and the beneath 4,1 mm or 5, a shelled from you for Fee, Machillen, New Ker, 1980, 5,51 Spare 2-21 Medice 4, Herbart, Kon, Operan, Toon Renor, Feedin, 1996, 1,1 Raper 2, 11 Raper 2, 11 Raper 2, 11 Raper 3, 11 R

In the lything has control and an admission of the control and an inflictibility of the lything has been admissible to the lything the lything and a lything the lything and a lything a lything and a lything and a lything and a lything and a lything ACTIONS

14.3 mm lare - version with power (e.g. -4.000; 0.007 mm) Pub. I are - version also power (e.g. -4.000; 0.018 mm) 8.4 mm 9.4 mm - 4.250; 0.009; 4.500; increments) +2.250; 0.009; 4.750; increments) +2.550; 0.009; 4.750; increments)

The ACLAULE DASYS® Brand Contact the following dimensions:

Diameter (DIA):

Center Thickness:

• On contractions was considered to the contraction of the contractio

The remainstrate and the contract departs to use displayer and red all outdoors are set for the sea of the contract and the contract departs to use of the contract departs and a fair to the set of the contract debar departs and a fair to the set of the contract between of it. Heart one address contracts the contract between of it. Heart one address contracts the contract between of it. Heart one of the contract

Always keep the bronse completely immersed in the recommended storage solution when Always keep the bronse completely work indiced. Provinged persists of large fig. as quoraging the lorer air for 30 minutes or morey will induce the adding of the lense surface to return to a wettable state. If the lense surface does become drived out, ducant the lense and use a new one.

The related and the state of the control of the con If type is Discuss with Pribates.

On the price of the pr

to demonstrate that wearing UV Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

In INJUST (STOP) and Continue in a chacked the dised current out of misches memoral proposal and legisters are the chacked the study of the charge of the ch

Lenese prescribed for therapeutic use may be worn for daily or extended

# GENERAL FITTING GUIDELINES

A remain execution

A format execution

Feltian indicate to war these innear should be closen launch on:

A fight in both an extra should be closen launch on:

• A fight is before installed and care for the benne

• A fight is controlled and care for the benne

• A fight is controlled and care for the benne

• A fight is controlled and care for the benne

• A fight is controlled and care for the benne

• A fight is controlled and care for the benne

• A fight is controlled and care for the benne

• A fight is controlled and care for the benne

• A fight is controlled and care for the probled with control force.

• A fight is controlled and care for the probled of the control for the parties of the control of the parties of the control of the parties of the control of the parties of the control of the parties of the control of the control of the control control of period and control of the cont

Board or this reduction, If it is determined that the patient is eligible to wear these because, the COLO Professional should proceed to the appropriate less titting in characters or effected between the color of the property than been titting in the color of the property of the property of the color of the property of the color of the property of the color of the property of the color of the property of the color of

exclusion designable and the state of the st

JJVC CONFIDENTIAL

When perceiping coutch less were the REPAUTING MLN When perceiping coutch less were the REPAUTING MLN When perceiping coutch less were the REPAUTING MLN WHITE ALSO A MLN WHITE A MLN WHIT

Coule institute to the capital making making with the capital that of countries in an experient is smooth, then the capital ca

nun wen.
FE PROBLEM, INCLIDING CORREAL LUCESS, DAN DEVELOP RAPDUY AND
LEAD TO LOSS OF WISION. IF THE PATIENT EXPERIENCES.
• The Processor of Annual Control

Other Ege Problems.

Other Ege Problems.

DI PROMET IN CONTACT THE ETC. CORE PROFESSORIAL.

DI PROMET IN CONTACT THE ETC. CORE PROFESSORIAL.

THE PROMET IN CONTACT THE ETC. CORE PROFESSORIAL.

THE REAL HE INTERCRETED OF IN SAME THE PROFESSORIAL.

THE REAL HE INTERCRETED OF IN

1. Others of a Encourt Fill term was a finish of the property of the processing of the processing in a finish of the the substant content to produce the content of the content of the content that and the processing of the processing of the processing of the processing of the the processing of th

If the sield loss care is japped to be let or sheep fitting, the alternate base care, analysis when the sield loss care is japped to be let or sheep fitting, the alternate has been districted by the less. The proper level is not if the common care is the site of the common care and the common care is the common care and care for the common care and care for the common care and care for the common care and care in the less of the common care and the less of the less 3. Others of a Steep Elling Lens.
A sheep fining lens may be the common of the Mouning characteristics result improvement with the blicks comparable infestions, and resistance when patients I hear up display with the lower list. If the lens is judged to be steep firms, it should be a selected.

# Alcon

# Package Insert for Alcon DAILIES TOTAL1™ for Astigmatism (delefilcon A) soft contact lenses for daily disposable wear

W900409251

PORTANT: This package insert is effective as of May 2020 and applicable to the deleticon A contact inness described below. Please read carefully and keep this information for future use is package insert is intended for the Tye Care Professional, but all doubt be made available to patients upon request. The Tye Care Professional study device the patient is intended for the Tye Care Professional study page to be stalled to the Tye Care Professional study page to be stalled to the Tye Care Professional study page to be stalled to the Tye Care Professional study page to the Tye Professional study page to the Tye Care Professional study page



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed Eye Care Professional.

### PRODUCT DESCRIPTION

DAILIES TOTAL 17th for Astigmatism (delefilicon A) soft contact lenses are made of a DAULES UNAL. "To Assignation (ceremon 4) soft contact tenses are made of a less material that is approximately 53% water and 57% (deleficon A) polymer, a silicone containing hydrings with added phosphatidy/icholine. The core lens material layer that exceeds 80% water. Lenses contain the color additive copyer phthatiogramine, and have a light blue-green tirt that makes them easier to see when handling. This package insert applies to DAULES TOTAL." We for adisparation lenses with light absorbing chromophores as identified in "Contents" statement on carbon handling. babeling). Bendiracele UV and UV-Vis absorbing monomers are used to block UV radiation and reduce transmittance of high energy visible light (HEVL) wavelengths in the range from 380 nm to 450 nm\*.

Lens Properties
• Refractive Index (hydrated): 1.42

 Light Transmittance:
 HEVL Transmittance: 90% ± 5% for average over 380 to 780 nm ≤ 80%T at 420 nm (refer to Figure 1 for

transmittance profile)\* τUVB < 1.0 % (average percent transmittance over 280 nm to 315 nm) I/V Transmittance

TUNA < 10.0 % (average percent transmittance over 315 mm to 380 nm) 140 barrer units, measured at 35 °C (intrinsic Dk -Coulometric method)

· Oxygen Permeability (Dk):

33% by weight in normal saline Water Content:

### Lens Parameters

Diameter Range: 13.0 to 15.0 mm -20.00 to +20.00 D Base Curve Range 8.0 to 9.2 mm

### DAILIES TOTAL 1<sup>TM</sup> for Astiomat m (delefilcon A)

Chord Diameter: 14.5 mm 0.11 mm @ -3.00 D (varies with power) Center Thickness

 Sohere Power: +4.00 to -6.00 D (0.25 D steps): -6.50 to -8.00 D

 Cylinder Power: -0.75 D, -1.25 D, -1.75 D, -2.25 D 10° to 180°, in 10° stens

When hydrated and placed on the comea, DAILIES TOTAL1™ for Astigmatism (delefficon A) soft contact lenses act as a refracting medium to focus light rays on

The lenses contain a combination of UV and UV-Vis blocking monomers to help The lenses contain a combination of UV and UV vis blocking monomers to help protect against transmission of narmal UV radiation to the comes and into the eye. For example, a lens with 0.09 mm center thickness (-3.00 D, thinnest projected parameter) blocks 37% of UVA radiation, and 99% UVB radiation average across the spectrum. The lenses reduce high energy visible light IVEVL, radiation reaching the back of the eye by about 33% in the range from 380 mm to 450 nm\*. See Figure 1 for the transmittance profile of detellion A lenses with light absorbing chromophores (-3.00 D, thinnest projected parameter). The radiation transmittance will be further control even the increase of the projected parameters. will be further reduced with increasing lens thickness

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV wanning or assorang contact lenses are NOT substitutes for protective UV absorbing eyewers, such as VM absorbing opgoler or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed. MOTEL Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental

cataracts. Exposure is based on a number of factors such as environmental conditions lathitude, eography, found overs) and personal factors (sethert and nature of outdoor activities). IV-Blocking contact lenses help provide protection against harmful IV radiation. However, clinical studies have not been done to demonstrate that wearing IV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. High energy visible light filtering provided by delettion A soft contact lenses with light absorbing chromophores is additive to the natural crystalline lens. There is no demonstrated clinical benefit to a 33% reduction in visible light at wavelengths below 450 nm. The Eye Care Professional should be consulted for more information.

Figure 1 illustrates the transmittance of a lens with 0.09 mm center thickness (-3.00 D, thinnest projected parameter), a human comea, a human lens, and the combined filtration effect of the contact lens and the human lens on retinal exposure. The shaded regions of the graph represent the integrated attenuation transmittance percentages of the defellion A lenses with light absorbing chromophores (-3.00 D, thinnest projected parameter) in the high energy visible light region (300 mm to 450 nm). The overall light attenuation over this region is 33%\*, with 65% attenuation over the region from 400 nm to 450 nm. This represents the filtration of the contact lens through the central 6 mm portion for a lens with 0.09 mm center thickness

(-3.00 D, thinnest projected parameter). Filtration would increase for contact lens powers with higher center thickness.

| Wavelength | Percent integrated attenuation<br>transmittance of high energy<br>visible light* |
|---|---|
| 380 nm to 400 nm | 85% |
| 400 nm to 450 nm | 21% |
| 380 nm to 450 nm | 33% |



- Delefilcon A with light absorbing chromophores: Contact lens with 0.09 mm center thickness measured through central 6 mm portion for the
- himset microless interaction of the man of the minimum of the mini
- Human crystalline lens from a 25 year old person as described in Waxler M., Hitchins V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida, 1986, p. 19, Figure 5.
- Combined filtering effect of the contact lens and the natural crystalline lens

on reunal exposure.

I've 1: Transmittance of a DAILIES TOTAL I<sup>TM</sup> for Astigmatism (delefike stact Lens versus a Human Cornea and a Human Crystalline Lens

INDICATIONS (Uses)
DAILES TOTAL 1<sup>TM</sup> for Astigmatism (deleticon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to 6.00 diopters (II) of astigmatism.

The lenses are to be used for single use, daily disposable wear (less than 24 hours while awake) only. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

### CONTRAINDICATIONS (Re

### DO NOT use delefilcon A soft contact lenses when any of the following exists:

- Inflammation or infection of the anterior chamber of the eve
- Any active disease, injury, or abnormality affecting the cornea, conjunctiva, or eyelids that may be exacerbated by contact lens wear
- Inadequate tear film (dry eye) that interferes with contact lens wear
- Reduced comeal sensitivity (comeal hypoesthesia)
- If eyes become red or irritated
- Use of any medication that is contraindicated or interferes with contact lens wear, including certain eye medications Any systemic disease which may be exacerbated by or interferes with safe
- contact lens wear, handling, or care
  Allergic reactions of the ocular surfaces or adnexa that may be caused by or
- exacerbated by the wearing of contact lenses
- Patient history of recurring eye or eyelid infections, adverse effects associated with contact lens wear, intolerance, or abnormal ocular response to contact lens

# Advise patients of the following warnings pertaining to contact lens wear:

- when paperess of the totolowing warnings portaining to contact lens wear: Problems with contact lenses and lens care products could result in serious injury to the eye. It is essential that patients follow their Eye Care Professional's directions and all labeling instructions for proper use of lenses and lens care products. Eye problems, including comeal ulcers, can develop rapidly and lead to loss of vision.
- It a patient experiences eye discomfort, foreign body sensation, excessive tearing, vision changes, or redness of the eye, the patient should be instructed to immediately remove lenses and promptly contact his or her Eye Care Professional. It is recommended that contact lens wearers see their Eye Care Professional regularly as directed.

  Studies have shown that contact lens wearers who smoke have a greater risk of suffering ulcerative keratifis than among those who are nonsmokers. <sup>2,1</sup>
- Daily week relative relative to the control whose the control of the control

- lenses overnight (outside the approved indication) compared to those who do not wear them overnight.

  Non-sterile liquids (i.e., tap water, distilled water, homemade saline solution, or
- saliva) should not be used as a substitute for any component in the lens care process. The use of tap and distilled water has been associated with Acanthamoeba keratitis, a comeal infection that is resistant to treatment and

### **PRECAUTIONS**

To prevent damage to the eyes or to the contact lenses, the folio precautions should be taken:

### Special Precautions for the Eve Care Professional

The following patients may not be suitable candidates and/or may experience a higher rate of adverse effects associated with contact lens wear:

- Patients with a history of non-compliance with contact lens care and disinfection regimen, wearing restrictions, wearing schedule or follow visit schedule.
- visit schedule.

  Patients who are unable or unwilling to understand or comply with any directions, warnings, precautions, or restrictions. Contributing factors may include but are not limited to age, infirmity, other mental or physical conditions, and adverse working or living conditions.

  Patients with diabetes may have reduced corneal sensitivity. As a result, they are more prone to corneal injury and will not heal as quickly or completely as non-diabetics.

Note regarding lens designs and parameters:

Due to the small number of patients enrolled in the clinical investigation of Due to the smail number of patients enrolled in the clinical investigation of lenses, all freship powers, design configurations, and lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, central and peripheral thickness, and optic zone diameter

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction. Therefore, the confining ocular health of the patient and less performance on the eye should be carefully evaluated on initial dispensing and monitored on an ongoing basis by the prescribing Eye Care Professional.

- bass by the prescribing Eye Care Professional.

  Note the following precautions during initial dispensing and subsequent visits:

  Fluorescein, a yellow dye, should not be used while the lenses are on the patient's eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used, the eyes should be flushed thoroughly with sterile saline solution that is recommended for in-eye use prior to inserting lenses. Avoid dispensing saline from an aerosol can directly into the eye.
- Instruct the patient to remove the lenses immediately if the eye becomes red or
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.
- Patients who wear contact lenses to correct prestyopia may not achieve the best corrected visual acuity for either far or near vision. Vision requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Before leaving the Eye Care Professional's office, patients should be able to promptly remove their lenses or should have someone else available who can remove their lenses for them.

# Eye Care Professionals should carefully instruct the patient to take the following care regimen and safety precautions:

- Be sure that before leaving the Eye Care Professional's office, the patient is able to promptly remove lenses or have someone else available to remove them. Good hygiene habits help promote safe and comfortable lens wear. Always wash, rinse, and dry hands with a lint-free towel before handling lenses.
- Intries, and cry names with a tractice error before beauting resource.

  Carefully follow the handling, insertion, removal, deaning, dininfecting, storing, and wearing instructions in the Patient Instruction Booklet for OAULES TOTALT<sup>IN</sup> for Assignatism (deleficion A) Soft Contact Lenses and any additional instruction. provided by the Eve Care Professional.
- Note the correct lens power for each eye to prevent getting them mixed up. Never use tweezers or other sharp objects such as fingemails to remove lenses from the lens container.
- Always handle lenses carefully. If a lens is dropped, small particles or fibers may adhere to the lens surface, which can irritate the eye. Replace with a sterile new
- . Discard any lens that has become dehydrated or damaged. Replace with a sterile

### Lens Wearing Precautions

- Remove the lenses before sleeping. Never exceed the prescribed wearing schedule regardless of how comfortable the lenses feel. Doing so may increase the risk of adverse effects.
- Always keep a supply of replacement lenses on hand or have back-up spectacles available, as lenses should not be reused. Do not share lenses with anyone as this may spread microorganisms, which could result in serious eye health problems.

- could read in sendors yet reading proceed.

  The lens should be disposed of each day upon removal from the eye.

  The lens should move freely on the eye at all times. If the lens sticks (stops moving) on the eye, follow the recommended directions in the CARE FOR A STICKING, TORK, DRY, OR DECENTERED LENS section. If non-movement of lens continues, consult your Eye Care Professional immediately.

<sup>\*</sup> See "Note". There is no demonstrated clinical benefit to a 33% reduction in visible light at wavelengths below 450 nm.

- · REMOVE THE LENS IMMEDIATELY if your eye becomes red or irritated
- Promptly remove the lens to avoid serious injury in the event that dust, a foreign body, or other contaminant gets between the lens and the eye.
- Avoid all harmful or imitating vapors and fumes while wearing lenses to reduce the chance of lens contamination or physical trauma to the eye.
- Eye irritation, infoction, or lens damage may result if cosmetics, lotion, seep, cream, hair spray, deodorant, aerosol products, or foreign particles come in contact with lenses. If sprays are used, eyes should be kept closed until the spray has extent.
- Growth an Eye Care Professional about wearing lenses during water sports and water related activities, Contact lens exposure to non-sterile water during activities such as swimming, water sking, and hot tube may increase the risk of ocular infection including, but not limited to, Azanthamoeta Neratilis.
- Never allow contact lenses to come into contact with non-sterile liquids (including tap water and saliva) as microbial contamination can occur, which may lead to permanent eve damage
- Do not use lenses beyond the expiration date.

### **Solution Precautions**

. Do not use saliva or any liquid other than the recommended solution for lubricating or rewetting drops with the lenses.

Other Topics to Discuss with Patients

- Periodic eye examinations are extremely important for contact lens wearers. Schedule and conduct appropriate follow-up examinations to determine ocula response. Alcon recommends that patients see their Eye Care Professional at least once each year or as recommended by the Eve Care Professional.
- near time clearly year on a recommend by the cyc during the retreased lens awareness, lens intolerance, blurred vision, or visional changes. These include, but are not limited to, antihistamines, decongestants, diuretics, muscle relaxants, tranquitizers, and those for motion sickness. Caution patients using these medications accordingly and prescribe proper remedial measures
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.

It is strongly recommended that patients be provided with a copy of the DAILIES TOTAL11\*\* for Astigmatism (deletiicon A) soft contact lens Patient instruction Book available from Alcon. It is important that patients understand its contents prior to

### Who Should Know the Patient is Wearing Contact Lenses

- Instruct patients to inform their employers that they are wearing contact lenses. Some jobs may require the use of eye protection equipment or may prohibit the wearing of contact lenses.
- instruct the patients to inform their health care professionals that they are wearing contact lenses, as certain medications may interfere with contact

### WATER ACTIVITIES

### Do not expose contact lenses to water while wearing them.

Water can harbor microorganisms that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when showering or swimming, discard them and replace with a new pair. Ask the Eye Care Professional for recommendations about wearing lenses during any activity involving water.

### ADVERSE EFFECTS (Possible Problems)

Patients should be instructed to check their eyes regularly to make sure they look well, feel comfortable, and vision is clear.

- Potentially serious complications are usually accompanied by one or more of the following signs and symptoms: Moderate to severe eye pain not relieved by removing the lens
- Feeling of something in the eye (foreign body sensation)
  Excessive watering or other eye secretions, including mucopurulent discharge
- · Redness of the eyes
- Sensitivity to light (photophobia
- · Burning, stinging, itching or other pain associated with the eyes
- t is less compared to when the lens was first placed on eye
- · Reduced sharpness of vision (poor visual acuity)
- · Feeling of dryness

These syr nptoms, if ignored, may lead to more serious complications.

### WHAT TO DO IF A PROBLEM OCCURS

If any of the above signs or symptoms occur:

• IMMEDIATELY REMOVE THE LENSES.

- . If the discomfort or problem stops, discard the lens and replace it with a new
- If the discomfort or problem continues after removing the lensies) or upon insertion of a new lens, IMMEDIATELY remove the lensies) and contact an Eye Care Professional for identification of the problem and prompt treatment to av serious eye damage.
- Eve Care Professionals should inform the patient that a serious condition such as coneal uice, uicerative keratifis, infection, comeal vascularization, or iritis may be present. These conditions may progress rapidly and may lead to permanent loss of vision. Less serious reactions such as brasions, infiltrates, and bacterial conjunctivitis must be managed and treated properly to avoid more serious
- complications.

  Additionally, contact lens wear may be associated with ocular changes that require consideration of discontinuation or restriction of wear. These include, but are not limited to, local or generalized conneal edema, epithelist microcysts, epithelist straining, infiltrate, provisorsalization, endothelial polymegathism, tarsal papillary changes, conjunctival injection, or iritis.

### CARE FOR A STICKING, TORN, DECENTERED, OR DRY LENS

Patients should be informed that it may be possible to resolve less serious problems associated with contact lens wear by following the directions below. However, if following these directions does not resolve the problem, patients should consult their

tollowing unless directions loves not exercise the processin, patients should crisis in Eye Care Professional immediately to avoid figury to the eye.

The lens should move freely on the eye at all times, if the lens sticks (stops moving) or begins to dry on the eye, apply several drops of a recommended lubricating solution (used in accordance with package labelling). Wait until the

lens begins to move freely on the eye before attempting to remove it. It is important that you wash and dry your hands thoroughly before removing the lens. If the lens continues to stick, IMMEDIATELY consult your Eye Care

- It a lens tears in your eye, remove the pieces carefully by pinching them as you would for normal lens removal. If the lens pieces do not seem to remove easily, do not pinch the eye tissue. Rilses with sailer. If this does not help, contact the Eye Care Professional for assistance.
- If a lens decenters on the eye, it may be possible to re-center it by:
  - o Closing your eyelids and gently massaging the lens into place, or
  - o Looking in the direction of the lens and blinking gently, or
  - Gently pushing the off-centered lens onto the comea with light finger pressure on the edge of the upper or lower eyelid.
- Occasional dryness may be relieved by blinking fully several times or by the use of contact lens rewetting drops that are approved for use with soft contact lenses. If dryness persists, consult your Eye Care Professional.

### **EMERGENCIES**

If chemicals of any kind (household products, gardening solutions, laboratory

- chemicals, dut.) are splashed into the eyes:

   Flush eyes immediately with fresh saline solution or tap water.

   Remove and discard lenses and immediately contact the Eye Care Professional or visit a hespital emergency room without delay.

### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of delefficon A contact lenses, please notify: Alcon Medical Affairs in the USA at

### FITTING GUIDE AND PATIENT ROOK! FT

Conventional methods of fitting contact lenses apply to DAILIES TOTAL1™ for Assignatism (oldeflicon A) contact lenses. For a detailed description of the fitting techniques, refer to the DALLES TOTAL. \*\* for Assignatism (oldeflicon A) soft contact lens Professional Etting and Information Guide for more information. Golder the Professional Etting and Information Guide and a Patient Instruction Booklet are lens Professional Fitting and Information Guide for m Professional Fitting and Information Guide and a Pat available free of charge from:

Alcon Laboratories, Inc.

Fort Worth, TX 76134-2099, USA

or by calling Alcon Customer Service in the USA at: 1-800-241-5999

### LENS WEAR AND REPLACEMENT SCHEDULE

- Daily Wear (less than 24 hours, while awake)
   Normal daily wear of lenses assumes a minimum of 6 hours of non-lens wear per 24-hour period; however, optimum individual wearing schedules will vary.
- The maximum daily wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition because individual responses to contact lenses vary.
- Daily wear patients may initially over-wear the lenses. Avoid this tendency by values was patients and an interference in the latest and the standards of stressing the importance of adhering to a proper initial wearing schedule. For patients who are new to daily wear, gradually increasing scheduled wearing time may allow ocular tissues to more easily adapt to contact lens wear.

### Lens Replacement

Deletition A contact lenses are intended to be worn once (daily disposable wear) and then discarded at the end of each wearing period. The patient should be instructed to start the next wearing period with a fresh new lens.

### LENS HANDLING INSTRUCTIONS

- Always wash and rinse hands thoroughly and dry completely with a clean, lint -free towel before handling contact lenses.
- Note the correct lens power for each eye to avoid getting them mix
- Do not use if blister package is damaged or not sealed completely. This may result in product contamination, which can lead to a serious eye infection.
- Shake the blister pack (containing a fresh new lens) gently prior to opening
- Remove the lens from the blister pack by carefully pouring it onto the palm of the
- Ensure that the lens is right side out.
- Inspect the lenses prior to insertion. Do not insert damaged or unclean lenses.
   Lens Insertion Instructions

- Wash and rinse hands thoroughly and dry completely with a clean lint-free
- Place a lens on the tip of your clean and dry right or left index finger. Place the middle finger of the same hand close to lower eyelashes and pull down the lower
- Use the fingers of the other hand to lift the upper eyelid.
- Place the lens directly on the eye (comea) and gently roll finger away from the
- Look down and slowly release the lower lid.
- Look straight ahead and slowly release the upper lid.

### Lens Removal Instructions

- Wash and rinse hands thoroughly, and dry completely with a clean, lint-free
- Blink fully several times.
- While looking up, use the tip of the finger to slide the lens down onto the white part of the eye.
- Remove the lens by pinching gently between thumb and forefinger. Do not pinch
- If the lens is difficult to grasp, dry fingers once more and try again. Do not use rewetting drops in this instance.
- Never use tweezers or other sharp objects such as fingernals to remove lenses from your eyes.
   LENS CARE DIRECTIONS

- To help avoid serious eye injury from contamination, the Eye Care Professional should review the following instructions with the patient:
   Cleaning and disinfection of daily disposable lenses is not recommended. The

patient should be reminded to have replacement lenses or back-up spectacles available at all times.

Do not use saliva, tap water, homemade saline solution, distilled water, or ng other than the recommended rewetting drops or lubricants indicated for

### DISPOSAL AND RECYCLING

Dispose of contact lenses and the blister pack lidding in the waste bin, not down th toilet or sink. The carton packaging and the polypropylene (PP) plastic shell of the blister pack should be placed in the waste bin or recycled according to local waste

Eye Care Professionals should educate contact liers technicians concerning proper use of thal lenses. Each contact liers is shopped sterile in a bitset peak containing proper use of thai lenses. Each contact liers is shopped sterile in a bitset peak containing properly subject of the proposition tenders should be throughly wested, rissed, and dried with a lint-free towel prior to handling a lens, in order to ensure sterility, the bitset peak should not be opened until immediately prior to use. For fitting and diagnostic purposes, the lenses should be disposed of after a single use and not be re-used from patient to patient.

### HOW SUPPLIED

Row SUPPLEU
Each lens is packaged in a foll-sealed plastic blister pack containing phosphate buffered saline solution with approximative) 0.3% of polymeric wetting agents consisting of copolymers of polymers and polylacrylamide-acrylic) acid and is steam stemized The package is marked with the base curve, diameter, dioptric power, cylinder racis and power (where applicable), ADD power (where applicable) manufacturing, and expiration date, Lenses are supplied in cartons containing up to 90 individually sealed contact lenses.

### The following may appear on labels or cartons:

| Symbol / Abbreviation | Description |
|---|---|
| BC | Base Curve |
| DIA | Diameter |
| PWR | Power |
| D | Diopter |
| L | Left |
| R | Right |
| CYL AXIS | Cylinder power and axis |
| UV | Ultra-violet |
| UVA | Ultra-violet A |
| UVB | Ultra-violet B |
| UV-Vis | Ultra-violet and Visible |
| HEVL | High Energy Visible Light (blue light) |
| 0 | Packaging waste license sign |
| 2 | Do not re-use |
| LOT | Batch code |
| ₽œ | Use-by date<br>(Expiry date) |
| 0 | Single sterile barrier system |
| PROPERTY. | Sterifized using steam |
| CE | European conformity mark |
| • | English (example of two letter code for the language) |
| Δ | Caution |
| | Consult instructions for use |
| (9) | Do not use if blister package is damaged |
| (8) | DO NOT DISPOSE LENSES IN TOILET OR SINK |
| | Manufacturer |
| اس | Date of manufacture |
| M2 | Medical device |
| == | Authorized representative in the European Community |
| (B) ordy | CAUTION: Federal (United States) law restricts this device<br>to sale by or on the order of a licensed eye care profession |

### Date: August 2021

Manufacturer: Alcon Laboratories, Inc. 6201 South Freeway Worth, TX 76134-2099, USA

<sup>1</sup> Check for actual product availability which may change over time.

<sup>2</sup> Outler GR, Chalmers RL, Roseman M. The Clinical Presentation, Prevalence, and Risk Factors of Focal Comeal Infiltrates in Soft Contact Lens Wearers. *The CLAO Journal*. Jan 1996: 22 (1): 30-37.

Schein OD, Glynn RJ, Poggio EC, Seddon JM, Kenyon KR. The Relative Risk of Ulcerative Keratitis Among Users of Daily-Wear and Extended-Wear Soft Contact Lenses The New England Journal of Medicine. 1989; 321(12):773-783.

### Alcon

© 2021 Alcon Inc.

W900409251-0821






































































































## Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

## PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6576 Evaluation of Lens Rotation in Habitual Wearers of Toric, Soft Contact Lenses

Version and Date: 1.0 03 October 2024

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155:2020¹, Declaration of Helsinki², United States (US) Code of Federal Regulations (CFR)³, and International Council for Harmonization Good Clinical Practice E6(R2) (ICH GCP)⁴ and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. I, as the Principal Investigator, am responsible for ensuring that all clinical site personnel, including Sub-Investigators, adhere to all regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial subjects.

All clinical site personnel involved in the conduct of this study will have completed Human Subjects Protection Training before participating in the study.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix H of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

| Principal<br>Investigator: | | |
|----------------------------|------------------------------------------|------|
| | Signature | Date |
| T 101 | Name and Professional Position (Printed) | |
| Institution/Site: | Institution/Site Name | |
| | Institution/Site Address | |